CLINICAL TRIAL: NCT00222300
Title: A Targeted Strengthening Program Following Total Hip Replacement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2002/01532
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-08-08 (Estimated); Status verified 2003-10

CONDITIONS: Total Hip Joint Replacement
Keywords: Total hip replacement; Strength training; Gait analysis

INTERVENTIONS:
Behavioral: Strength training program

SUMMARY:
Total Hip Replacement (THR) is a common surgical procedure performed in people with hip osteoarthritis and appears to be effective in relieving pain and improving function. However significant wasting and weakness of the hip and knee muscles persists post-operatively. Although relief of pain and improvement of function are important outcomes following THR, weakness of the hip and knee muscles reduces a person's ability to manage stairs, slopes, public transport and results in persistent gait abnormalities. Since lower limb weakness is one of the risk factors for falls, it is important that patients undergo a strengthening program post-operatively. The hypothesis is that lower limb strength and function will be better in patients who undergo a strengthening program post-operatively than in those who have usual care.

DETAILED DESCRIPTION:
Total Hip Replacement (THR) is a common surgical procedure performed in people with hip osteoarthritis and appears to be effective in relieving pain and improving function. However significant quadriceps atrophy and weakness persist post-operatively. Although relief of pain and improvement of function are important outcomes following THR, weakness of the hip and knee muscles reduces a person's ability to manage stairs, slopes, public transport and results in persistent gait abnormalities. Since lower limb weakness is one of the risk factors for falls, it is important that this is appropriately addressed.

The study examines the effect of an eight-week task-specific strengthening program on lower limb function in patients following THR in a randomized controlled trial. The experimental program is being conducted as a circuit in a gymnasium environment. Changes on specific measures of physical function of patients in the Experimental Group will be compared with those of patients in a Control Group who will continue with the standard care program provided at Austin Health.

Outcome measures include:lower limb muscle strength using a step test, pain, stiffness, and function as reported on the WOMAC questionnaire, quality of life using the AQoL questionnaire, the Timed Up-and-Go test. Walking tests will also be conducted. These include:

1. Walking pattern, recorded on an instrumented mat
2. Walking endurance measured by the 6-minute walk test.
3. Analysis of hip joint torques using 3-D motion analysis.

ELIGIBILITY:
Inclusion Criteria:

* primary uncomplicated total hip joint replacement 6-8 weeks prior to enrolment.
* able to walk 45m independently with or without walking aid.
* able to comprehend instructions
* prior joint replacement on the other side at least 12 months previously

Exclusion Criteria:

* unable to fully weight-bear on affected limb
* pre-existing neurological or orthopaedic condition affecting gait
* revision surgery
* post-operative complications, e.g. wound infection
* uncontrolled systemic disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-05; Study Completion 2005-12

PRIMARY OUTCOMES:
Lower limb strength using a step test

SECONDARY OUTCOMES:
Pain, stiffness and function using the WOMAC questionnaire.
Function using the Timed Up-and-Go Test.
Quality of life using the AQoL
Spatiotemporal measures of walking using an instrumented mat.
Hip joint torques using 3-D motion analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Galea, PhD, Principal Investigator — University of Melbourne
Locations (1):
- Austin Health, Melbourne, Victoria, Australia